CLINICAL TRIAL: NCT04713072
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding Clinical Trial in Patients With Active Psoriatic Arthritis to Investigate Efficacy, Tolerability, Safety, Pharmacokinetics and Immunogenicity of ABY-035
Brief Title: A Study to Investigate Efficacy, Tolerability and Safety of ABY-035 in Patients With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABY-035-202
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-11

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABY-035 40 mg (Experimental): 40 mg ABY-035 SC
  Interventions: Biological: ABY-035
- ABY-035 80 mg (Experimental): 80 mg ABY-035 SC
  Interventions: Biological: ABY-035
- Placebo (Placebo Comparator): Placebo, switching to 80 mg ABY-035 after 16 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ABY-035 — ABY-035 solution for injection
  Arms: ABY-035 40 mg; ABY-035 80 mg
Biological: Placebo — Placebo to ABY-035 solution for injection
  Arms: Placebo

SUMMARY:
This is a Phase II, prospective, multicenter, randomized, double-blind, placebo-controlled, dose finding trial in parallel-groups with primary endpoint at Week 16 (visit V9) to investigate the efficacy, tolerability, safety, pharmacokinetics and immunogenicity of ABY-035 in adult patients with PsA.

DETAILED DESCRIPTION:
The study evaluates two dose levels of ABY-035, in comparison to placebo, in subjects with psoriatic arthritis. The clinical trial duration is 72 weeks (Screening - last FU visit) comprised of up to 4 weeks of screening, 44 weeks of double-blind-treatment, and 24 weeks of follow-up.

Treatment Periods are:

* Treatment Period I: from V1 (Week 0) to V9 (Week 16)
* Treatment Period II: from V9 (Week 16) to V16 (Week 44: last dosing)

At visit V1 (Week 0), patients who meet the entry criteria will be randomly assigned in equal rates (1:1:1) to one of three parallel groups (A, B, C).

The treatment will be administered once every 2 weeks (Q2W).

Patients assigned to groups A and B will receive active treatment from V1 to V16 (group A = 40 mg ABY-035; group B = 80 mg ABY-035). Patients initially assigned to placebo will switch to active treatment at visit V9 in a blinded fashion (group C = Placebo from V1 to V8 and 80 mg ABY-035 from V9 to V16).

ELIGIBILITY:
Inclusion criteria:

* Patient who has given his / her signed declaration of consent and data protection declaration
* At least 18 years and less than 75 years of age at Screening visit
* Psoriatic arthritis with inflammatory musculoskeletal disease (joint, spine, or entheseal) with the presence of ≥3 points from the five categories of the Classification Criteria for Psoriatic Arthritis (CASPAR) at any timepoint in medical history.
* Active psoriatic arthritis defined by:
* ≥3 swollen joints out of 66 joints (SJC66) at Screening visit and Baseline visit
* ≥3 tender joints out of 68 (TJC68) at Screening visit and Baseline visit
* Precedent failure or insufficient treatment response to or contraindication or intolerability to nonsteroidal anti-inflammatory drug (NSAID), csDMARD (i.e. MTX, sulfasalazine, leflunomide, hydroxychloroquine, cyclosporine A), and/or TNFi (e.g. adalimumab, infliximab, etanercept, golimumab, certolizumab)
* Rheumatoid factor (RF) and anti-CCP antibody negative
* Presence or history of plaque psoriasis

Exclusion Criteria:

* Underlying conditions which significantly immunocompromise the patient and / or place the patient at unacceptable risk for receiving an immunomodulatory therapy
* History of or current relevant autoimmune diseases (e.g. rheumatoid arthritis, primary ankylosing spondylitis, systemic lupus erythematosus) other than psoriasis or psoriatic arthritis
* History of or current fibromyalgia or pain syndrome
* Uncontrolled inflammatory bowel disease
* Presence or history of recurrent or medically important infections in the last 6 months prior to Baseline visit
* Clinically relevant Candida infection requiring systemic treatment within the last 6 months prior to Baseline visit
* History or any signs of lymphoproliferative disease, or a known malignancy or a history of malignancy within the previous 5 years
* Insufficiently controlled heart failure
* Current uncontrolled arterial hyper- or hypotension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 50 response rate (ACR50) | 16 weeks
  ACR50 response rate at V9 (Week 16) for higher Dose vs. Placebo
ACR50 | 12 weeks
  ACR50 response rate at V7 (Week 12) for higher Dose vs. Placebo

SECONDARY OUTCOMES:
ACR20/70 | 16 weeks
  ACR20/70 response rate, percentage of patients achieving Minimal Disease Activity (MDA): at V9 (Week 16) for higher Dose vs. Placebo
ACR20/70 | 12 weeks
  ACR20/70 response rate, percentage of patients achieving MDA: at V7 (Week 12) for higher Dose vs. Placebo
ACR20/50/70 | 16 weeks
  ACR20/50/70 response rate, percentage of patients achieving MDA: at V9 (Week 16) for Lower Dose vs. Placebo
ACR20/50/70 | 12 weeks
  ACR20/50/70 response rate, percentage of patients achieving MDA: at V7 (Week 12) for Lower Dose vs. Placebo
ACR 20/50/70 | 8 weeks
  ACR 20/50/70 response rate, percentage of patients achieving MDA: at V5 (Week 8) for higher Dose vs. Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Myreen Tomas, MD, Study Director — ACELYRIN Inc.
Locations (32):
- Austria (3):
  - LKH-Univ. Klinikum Graz Universitätsklinik für Innere Medizin Klinische Abteilung für Rheumatologie und Immunologie, Graz
  - Medizinische Universität Innsbruck/Tirol Kliniken GmbH Universitätsklinik für Innere Medizin II, Innsbruck
  - Vienna Medical University Department of Internal Medicine III Division of Rheumatology, Vienna
- Katholieke Universiteit Leuven, Leuven, Belgium
- Czechia (4):
  - VESALION s.r.o., Ostrava
  - Revmatologický ústav, Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - PV Medical Services s.r.o., Zlín
- Germany (7):
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Schlosspark Klinik, Berlin
  - Centrum für Innovative Diagnostik und Therapie Rheumatologie/Immunologie, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Rheumazentrum Ruhrgebiet Herne, Herne
  - Klinikum der Universität München Rheumatologie, München
  - Rheumazentrum Ratingen, Ratingen
- Hungary (4):
  - Qualiclinic Kft., Budapest
  - CRU Hungary Ltd, Miskolc
  - MÁV Kórház és Rendelőintézet, Reumtólegia, Szolnok
  - Vital Medical Center, Veszprém
- Poland (7):
  - Nasz Lekarz Ośrodek Badań Klinicznych, Bydgoszcz
  - PRATIA MCM Krakow, Krakow
  - Centrum Medyczne AMED oddział w Łodzi, Lodz
  - ETYKA Ośrodek Badań Klinicznych, Olsztyn
  - ETG Skierniewice, Skierniewice
  - ETG Warszawa, Warsaw
  - Centrum Medyczne AMED, Warsaw
- Spain (6):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario Reina Sofía 1 Planta Derecha Servicio Reumatología- IMIBIC, Córdoba
  - Cliníca Ceta - Unidad de Ensayos Clínicos, Madrid
  - Hospital Parc Tauli de Sabadell, Sabadell
  - Complejo Hospitalario Universitario de Santiago de Compostela Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Quironsalud Infanta Luisa Unidad De Investigación De Reumatología, Seville

IPD SHARING:
Plan to Share IPD: No